CLINICAL TRIAL: NCT00636662
Title: Evaluation of the RAMP FLU A+B Test Versus Viral Culture Using Clinical Nasal Swab Samples From Patients With Suspected Influenza Infections
Brief Title: FLU A+B Nasal Swab Clinical Study
Acronym: FLUA+B
Status: Completed | Type: Observational
Sponsor: Response Biomedical Corp. (Industry)
Responsible Party: Sponsor
Other Study IDs: CSP012
Record Dates: First submitted 2008-03-07; First posted 2008-03-14 (Estimated); Last update posted 2019-03-27 (Actual); Status verified 2019-03

CONDITIONS: Influenza
MeSH Terms: conditions — Influenza, Human

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — mucous
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- all: any patient exhibiting symptoms of influenza
  Interventions: Other: Non-invasive diagnostic testing

INTERVENTIONS:
Other: Non-invasive diagnostic testing — No patient treatment is altered by enrollment in this trial

SUMMARY:
The purpose of this clinical study is to obtain clearance for the nasal swab sample type by demonstrating the performance characteristics of the FLU A+B Test versus standard laboratory culture for Influenza A and B viruses using nasal swab samples.

DETAILED DESCRIPTION:
Patients exhibiting symptoms of influenza enrolled in a fashion that confidentiality of all personal health information is maintained.

No patient treatment is affected by enrollment in this trial.

ELIGIBILITY:
Inclusion Criteria:

* Male and Female of all age groups
* Patients exhibiting influenza symptoms (i.e., fever, body aches, headaches, cough, sore throat, and other respiratory symptoms) at the time of examination
* Patients must either present with a fever (>100ºF; >37.8ºC) at time of examination or have had a fever (>100ºF; >37.8ºC) or declare at time of the examination that they had a fever within the previous 3 days prior to the examination
* Must be able to collect sample using the nasal swab sample type

Exclusion Criteria:

* Patients with no fever at time of examination or within the 3 days prior to examination and/or are currently undergoing treatment (including anti-virals) will be excluded from the study.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Nasal swab samples will be collected from subjects suspected of having influenza infections and onset has occurred within 3 days of examination. Across the sites these samples will be drawn from an approximately 60% pediatric patients (<21 years), and 40% adult patients (>21 years) and it is expected that the population will be divided approximately equally between males and females.
Sampling Method: Non-Probability Sample
Enrollment: 800 (Actual)
Dates: Start 2008-02; Primary Completion 2008-05 (Actual); Study Completion 2008-05 (Actual)

PRIMARY OUTCOMES:
Support the addition of nasal swab sample type to labeling for the FLU A+B Test. The nasal swab sample data will be analyzed for the FLU A+B Test versus standard laboratory culture identification to determine the sensitivity and specificity. | 1 day

CONTACTS AND LOCATIONS:
Locations (5):
- United States (4):
  - Northwestern University, Chicago, Illinois
  - Washington University / St. Louis Children's Hospital, St Louis, Missouri
  - Wake Forest University Health Sciences, Winston-Salem, North Carolina
  - Dell Children's Hospital, Austin, Texas
- Mt. Sinai Hospital, Toronto, Ontario, Canada